CLINICAL TRIAL: NCT06497595
Title: Exercise and Nutritional Intervention to Reduce the Risk of Sarcopenia in Older Adults With Type 2 Diabetes and Obesity Treated With Semaglutide: A Randomized Controlled Trial
Brief Title: Lifestyle Intervention to Reduce the Risk of Sarcopenia in Adults With Diabetes & Obesity Treated With Semaglutide
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Dr. Tali Cukierman-Yaffe, professor, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1072-24-SMC
Record Dates: First submitted 2024-06-27; First posted 2024-07-12 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Type 2 Diabetes Mellitus in Obese
Keywords: older adults; sarcopenia; obesity; type 2 diabetes; semaglutide; exercise; physical capacity
MeSH Terms: conditions — Sarcopenia; Obesity; Diabetes Mellitus, Type 2; Motor Activity | interventions — semaglutide; Exercise; Nutritional Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- multi-disciplinary intervention group (MDIG) (Experimental): Participants in this group will receive Semaglutide 2.4 mg SC QW and take part in a multi-disciplinary intervention comprised of home-based exercise and nutritional counselling for the 26-week trial duration.
  Interventions: Behavioral: Wegovy (2.4 Mg Dose) + exercise & nutrition
- general health recommendations control group (GHRG) (Active Comparator): Participants in this group will receive Semaglutide 2.4 mg SC QW and general health recommendations for the 26-week trial duration.
  Interventions: Other: Wegovy (2.4 Mg Dose) + usual care

INTERVENTIONS:
Behavioral: Wegovy (2.4 Mg Dose) + exercise & nutrition — Participants will participate in a 26-week, tri-weekly, exercise program. One 45-minute exercise session will be provided via a virtual meeting platform each week and recorded. The participants will be asked to independently repeat each recorded session twice on separate, non-consecutive days of the week without supervision. The program will focus on progressive resistance exercises using body weight, a resistance band and various household items. A weekly follow-up call will be conducted to gather feedback and monitor adherence along with a personal exercise diary that each participant will fill out and bring to each on-site visit. Each exercise session will be performed in small groups and will be administered by a fitness specialist. In addition, participants will receive personal individualized nutritional counseling which will be administered every 2-4 weeks online via ZOOM. A certified dietitian will conduct all diet sessions.
  Arms: multi-disciplinary intervention group (MDIG)
Other: Wegovy (2.4 Mg Dose) + usual care — Participants will receive dietary guidance as customary among patients with type 2 diabetes (T2D) and obesity monitored in a diabetes clinic. Additionally, general recommendations for physical activity (PA) according to the medical guidelines for PA for T2D will be given. Guidelines recommend 150 minutes or more of moderate to vigorous-intensity aerobic activity per week, spread over at least 3 days/week, with no more than 2 consecutive days without activity, or engage in 75 minutes/week of vigorous-intensity or interval training (for more physically fit individuals). Incorporate 2-3 sessions/week of resistance exercise on nonconsecutive days, decrease sedentary behavior and add flexibility and balance training 2-3 times/week. Participants in the GHRG will be requested to fill out an exercise diary (report on unsupervised training days) and a 2-day food diary for periodic monitoring which they will bring with them to each on-site visit.
  Arms: general health recommendations control group (GHRG)

SUMMARY:
This study aims to test whether a multi-disciplinary intervention involving exercise and nutrition can slow down the decline in physical function, muscle strength and mass in older adults (aged 65-75) with Type 2 diabetes (T2D) and obesity treated with Semaglutide.

The main questions it aims to answer are:

In older people with T2D and obesity, treated with Semaglutide, does a multi-disciplinary intervention of exercise and nutrition compared to standard health recommendations:

1. Reduce the rate of decline in muscle mass?
2. Reduce the rate of decline in muscle strength?
3. Reduce the rate of decline in physical function?

Participants will:

Administer Semaglutide once weekly for 6 months. Visit the clinic once every 8 weeks for checkups and tests. Keep a diary of their exercise and food consumption. Participants in the intervention group will participate in an online exercise program and will receive personal nutritional counseling.

DETAILED DESCRIPTION:
The study will be conducted at the Center for Successful Aging with Diabetes, Sheba Medical Center and the Clinical Research Center for Diabetes, Hadassah Medical Center, Israel. The research will include a team with expertise in endocrinology, nutritional interventions, physical therapy, fitness training, medical imaging and biostatistics.

Participants aged 65-75 years, with both type 2 diabetes (T2D) and overweight / obesity, will be randomly allocated to either a (1) Semaglutide and multi-disciplinary intervention group (MDIG) comprised of exercise and diet or (2) Semaglutide and general health recommendations control group (GHRG). The drug dosage (Wegovy, Semaglutide) will be gradually increased every 4 weeks starting with 0.25 milligrams (mg) on week 0 and reaching 2.4 mg by week 16 as per the Wegovy label and maintained at 2.4 mg until the end of the trial (week 26). If a participant is unable to tolerate the 2.4 mg subcutaneous weekly dose (SC QW) of Semaglutide, the highest tolerable dose will be administered, with continued efforts to gradually increase the dose over time.

Participants in the MDIG will undergo a once-weekly group exercise training that will be delivered online, followed by 2 unsupervised home-based sessions. Weekly phone calls and a personal exercise diary will be used in order to measure adherence to the exercise program. In addition, personal nutritional counseling will be administered by a certified dietitian every 2 weeks for the first 4 weeks and every 4 weeks for the remaining 22 weeks via a virtual meeting platform (i.e., "ZOOM"). In addition, a 2-day food diary will be filled out for tracking and documentation. All group exercise training will be conducted via a virtual meeting platform as well. Participants allocated to the GHRG will receive general health recommendations both verbally and in writing and continue with their regular daily routine. They will also be required to complete a personal exercise and food diary.

Visit 1- screening: All potential eligible subjects will be invited for a screening Visit, during which the following information would be obtained: a) Informed consent; b) Eligibility criteria form; c) Physician interview and examination; d) Demographic and medical information; e) Medical History and recent blood work.

Visits 2 - 5: After being allocated to the two study arms, 4 additional measurement visits will be booked: (1) baseline - week 0 (visit 2), (2) week 8 (visit 3), (3) week 16 (visit 4), and (4) end of treatment - week 26 (visit 5). The following information will be collected on each visit: a) Anthropometric measurements, including waist and hip circumference, waist to hip ratio, weight, height and body mass index (BMI, calculated in kg/m2); b) Body composition measured with Magnetic Resonance Imaging (MRI) and Dual-energy X-ray Absorptiometry (DXA); c) Functional and strength assessments, including balance, aerobic capacity, gait speed and strength tests d) Blood pressure (BP) and heart rate (HR) e) lipid profile and hemoglobin A1C test (HbA1C) (only on visits 2 and 5); f) frailty assessment (only on visits 2 and 5); g) Distribution of Semaglutide, usage and titration guidance (only visits 2-4) ; h) Documentation of 2-day self-reported food diary for MDIG (only on visits 3-5) i) Nutritional counseling for MDIG; j)collection and recording of partly used and full pens for estimation of Semaglutide adherence (only on visits 3-5); k) Documentation of exercise adherence through self-reported exercise diary (only on visits 3-5); l) Target Physical Examination; m) Adverse events collection (only on visits 3-5). All baseline measurements will be conducted within one week before the trial commences.

Measures of compliance/adherence: Compliance to the drug would be monitored in both arms. Consumption of <80% or >120% of study background medication (Semaglutide) would be considered poor adherence to therapy. Patients will be instructed to bring back all empty, partly used and full Semaglutide pens at each site visit and all pens will be counted and estimation of Semaglutide adherent will be recorded. In the MDIG, the subject's adherence to the exercise regimen will be assessed during weekly phone calls based on subject reporting and by documentation in a personal diary they will bring to each visit. Good compliance/adherence would be considered as performing ≥ 2 of the exercise sessions. In order to perform a protein consumption evaluation, the nutritional sessions will be recorded, and the patients will be asked to fill out a 2-day food diary before each visit.

Glucagon-like Peptide-1 Receptor Agonist (GLP-1-RA) treatment: All patients will receive Semaglutide 2.4 mg once a week for 26 weeks. Semaglutide will start at 0.25 mg per week and escalate in a fixed-dose regimen every 4 weeks until the target dose is reached (i.e., 2.4 mg by week 16 until the end of trial). If a participant will not be able to tolerate Semaglutide 2.4 mg SC QW dose, the highest tolerable dose of Semaglutide will be used and further attempts to increase Semaglutide dose will continue.

Changes in body composition will be carried out using whole-body MRI, DXA and body composition measures.

Functional assessments will include the following tests:

1. Timed up and Go (TUG) test which examines dynamic balance and mobility skills. The participant is asked to get up from a chair with handles, walk three meters, turn, walk back, and sit down in the shortest possible time. Data suggests that the TUG test is a reliable and valid test for quantifying functional mobility and risk for falls that may also be useful in following clinical change over time.
2. Short Physical Performance Battery (SPPB): The SPPB is an objective assessment tool for evaluating three domains of lower extremity physical function in older adults: balance, repeated chair stands, and gait speed. It is associated with various adverse health outcomes in older adults, including mobility impairments, difficulties performing basic activities of daily living (ADL) or instrumental activities of daily living (IADL), and falls. Poor performance on the SPPB and its components independently predict higher fall risk over 1 and 4 years of follow-up.
3. The 6-minute walk test (6MWT). The 6MWT assesses aerobic capacity. The test measures the distance walked over six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The 6MWT has been linked to frailty and mortality in older adults.

4.10-meter walk (10MW): The 10MW determines gait speed. The participant is asked to walk at a "comfortable pace" for 14 meters. The score achieved is determined by the walking time of the central 10 meters. Studies have shown that better gait speed is associated with a lower risk for functional decline, hospitalization and mortality.

Strength tests:

1. 30 second chair stand (STS): The purpose of this test is to evaluate lower limb muscle strength. The instructions are to get up from sitting to standing as many times as possible without the assistance of the arms for 30 seconds. The number of times within 30 seconds that the participant succeeds to rise from a seated position is counted. The strength of the lower limb muscles has a crucial impact on daily function. Failure to perform STS movements efficiently and smoothly may lead to falls.
2. Hand grip strength test: The maximum grip strength test evaluates upper limb strength using the Jamar dynamometer. The test is conducted in a neutral hand position and repeated 3 times. Grip strength assessment has been shown to have predictive validity and low values are associated with falls, disability, impaired health-related quality of life and prolonged length of stay in hospital as well as increased mortality.

Screening for frailty will be performed using the Fried scale. The scale includes five criteria, and pre-frailty is defined as the presence of two components while frailty is defined as the presence of at least three of the following components: (1) unintentional weight loss - loss of 10 lbs/4.5 kg or more in 1 year; (2) self-reported exhaustion / fatigue; (3) low physical activity level as assessed by a modified Baecke questionnaire; (4) slow gait speed - less than 0.8 m/s with or without a walking aid; (5) low grip strength relative to gender and body weight.

Anthropometric measurements: Weight and height, with body mass index (BMI) calculated as kg/m2 and waist and hip circumference measured, and waist to hip ratio calculated.

Glycemic control (GC): Hba1c will be collected at baseline and at the end of trial.

Socio-demographic questionnaire: Socio-demographic characteristics, including age, gender, education, marital status, employment status, ethnicity, and smoking status, will be collected at visit 1.

Discontinuation: Participants may withdraw consent for any reason at any time or be discontinued from the trial by the investigator if, based upon his clinical judgment, continuation in the trial is deemed inappropriate. In addition, the investigator may discontinue a subject if enrollment into the trial is inappropriate, the trial plan is violated, or for administrative and/or any other safety reasons or if the trial is terminated early for any reason.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 65-75 years old.
2. Patients who were previously diagnosed with type 2 diabetes.
3. Overweight / obesity (body mass index, BMI ≥ 27 kg/m2).

Exclusion Criteria:

1. Patients with significant hearing or visual disability.
2. Patients with Estimated Glomerular Filtration Rate (eGFR)<30 ml/min/1.73 m2.
3. Patients who are in active nutritional therapy.
4. Patients who changed their diet recently (< 1 month) and/or in a weight-loss program with >5% weight loss or used anti-obesity drugs in the last 3 months.
5. Patients who reported a weight loss of >5kg within 90 days of screening
6. Patients who were on Glucagon-like peptide-1 receptor agonists (GLP-1-RA) treatment during the last 3 months.
7. Patients with musculoskeletal disorders, which, by the judgment of the investigators, would limit their ability to perform the exercise training.
8. Patients with neurological diseases, which by the judgment of the investigators, would affect their ability to participate in the trial.
9. Patients with a history of amputation that impairs their ability to participate in the exercise program.
10. Patients with disabilities, which, by the judgment of the investigators, would affect their ability to participate in the trial.
11. Patients who use a walking aid.
12. Patients who are currently using systemic steroids.
13. Patients with active oncological diseases, excluding non-melanoma skin cancer.
14. Patients with diagnosed dementia or cognitive impairment that, in the view of the researchers, may impair their ability to sign a consent form or participate in the trial.
15. Patients who were hospitalized in the past month.
16. Patients who exercise regularly and in the eyes of the examiner will not benefit from the intervention program.
17. Anyone who is not suitable to participate in the study, according to the researcher's discretion.
18. Any contraindication to Magnetic resonance imaging (MRI) (e.g., MRI non-compatible cardiac implantable electronic device, metallic foreign bodies, implantable neurostimulation system, cochlear implants/ear implant, non-removable drug infusion pumps, catheters with metallic components, cerebral artery aneurysm clips which), or inability to perform an MRI scanner (e.g., claustrophobia).
19. Patients who do not fit within the measurement field of view of the Dual-energy X-ray absorptiometry (DXA) scanner in a supine position with the arms next to the body.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-30 (Estimated); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Thigh muscle volume (TMV) | 26 weeks
  Change in TMV from baseline to week 26

SECONDARY OUTCOMES:
Thigh muscle volume (TMV) | 26 weeks
  TMV value in week 26
Sit to stand test (STS) score | 26 weeks
  Absolute and relative change in Sit to stanf test score from baseline to week 26. The number of times the participant stands up and sits down from a chair within 30 seconds is measured. The test results are compared to norms according to the participant's age and gender to assess lower limb strength. The higher the number of repetitions, the better the lower limb strength.
Hand grip strength test score | 26 weeks
  Absolute and relative change in hand grip measurement from baseline to week 26. The subject is instructed to squeeze the hand dynamometer with maximum isometric effort, which is maintained for about 5 seconds. The test results are compared to norms according to the participant's age and gender to assess upper limb strength. A score < 27 kg for men and < 16 kg for women is considered a risk for sarcopenia.
Timed up and go (TUG) test score | 26 weeks
  Absolute and relative change in Timed up and go test score from baseline to week 26. The time it takes the participant to rise from a chair, walk 3 meters and return to a seated position is measured. The test results are compared to norms according to the participant's age and gender to assess dynamic balance and fall risk. The shorter the time taken to complete the task, the higher the ability, with a result over 14 seconds indicating an increased risk of falls.
6-minute walk test (6MWT) score | 26 weeks
  Absolute and relative change in the 6-minute walk test score from baseline to week 26. The distance covered over 6 minutes is used as the outcome by which to compare changes in performance capacity. The test results are compared to norms according to the participant's age and gender to assess aerobic capacity and endurance. A longer distance covered indicates better aerobic capacity and physical performance.
10-meter walk test (10MWT) score | 26 weeks
  Absolute and relative change in the 10-meter walk test score from baseline to week 26. The time it takes the participant to walk at a comfortable pace for 10 meters is measured. A score ≤ 0.8 meter per second (m/s) indicates low physical function and risk for falls.
Short physical performance battery (SPPB) test score | 26 weeks
  Absolute and relative change in the SPPB test score from baseline to week 26. The test includes three different domains (walking, sit-to-stand and balance) to assess functional mobility. The total score ranges from 0-12, a high score indicates high functional capacity while a score below 8 indicates low functional capacity and raises the suspicion of sarcopenia.
Fried Frailty scale | 26 weeks
  Change in state of frailty from baseline to week 26. The fried frailty scale includes five components, unintentional weight loss (10 lbs. in the past year), self-reported exhaustion, weakness (grip strength), slow walking speed, and low physical activity. The presence of one or two deficits indicates pre-frailty, and a total of three or more deficits indicate frailty, while the absence of deficits indicates a robust state.
Fat distribution | 26 weeks
  Absolute and relative change in total fat mass from baseline to week 26
Total lean mass | 26 weeks
  Absolute and relative change in total lean mass from baseline to week 26
Appendicular lean mass | 26 weeks
  Absolute and relative change in appendicular lean mass from baseline to week 26
Muscle quality (muscle fat infiltration) | 26 weeks
  Absolute and relative change in muscle fat infiltration from baseline to week 26

CONTACTS AND LOCATIONS:
Overall Officials: Tali Cukierman - Yaffe, professor, Principal Investigator — Division of Endocrinology, Sheba Medical Center, Israel.
Locations (2):
- Israel (2):
  - Hadassah Medical Center, Jerusalem
  - Sheba medical center, Ramat Gan